CLINICAL TRIAL: NCT03935165
Title: Indocyanine Green and Near-Infrared Vision in Deep Infiltrating Endometriosis Surgery. A Prospective Study (GRE-Endo-2 Trial)
Brief Title: Prospective Evaluation of Near-infrared Fluorescence Imaging Use as a Supportive Tool in Deep Infiltrating Endometriosis Surgery
Acronym: GRE-Endo-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Head of Department of Women's and Children's Health, Policlinico Agostino Gemelli Foundation University Hospital, Rome, Italy, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 736513. A 287 / C.E./2013
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Pelvic Endometriosis; Endometriosis Outside Pelvis
Keywords: indocyanine Green; deep Infiltrating Endometriosis; near-Infrared Vision; occult endometriosis; invisible endometriosis
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: In the selected patients, after a first white light visual inspection, 0.25 mg/(kg BW) ICG were injected intravenously. After 15 to 30 minutes a second inspection of the abdomen and pelvis in Near Infrared vision was made. All the visualized lesions were carefully described pre and post the Indocyanine Green injection, removed and listed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indocyanine Green arm (Experimental): All the patients to be enrolled have to meet the inclusion criteria. All enrolled patient is subjected, during laparoscopy, to an accurate inspection of the abdomen and all the visible endometriotic lesions are described.
  Subsequently, 0.25 mg /(kg BW) Indocyanine Green is administered intravenously during surgery and a second look of the abdomen and pelvis with the Near Infrared Vision is made, in order to identify the fluorescent lesions. All the lesions are described and localized pre and post the Indocyanine Green injection and then removed and properly cataloged.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — 0.25 mg /(kg BW) Indocyanine Green PULSION®/ VERDYE Diagnostic Green®
  - Indocyanine Green is administered Intravenously

SUMMARY:
The aim of the study is to establish a new and more accurate method to visualize the peritoneal changes caused by endometriosis using Indocyanine Green mediated fluorescence imaging. The hypothesis is that Indocyanine Green, a fluorescent dye that has wide applications throughout medicine in identifying vascularity of tissues and neo-vascularization, could facilitate the localization and excision of endometriotic lesions exploiting the hypervascularization due to the chronic inflammation. The already published Pilot Study GRE-ENDO (Cosentino F, Near-Infrared Imaging with Indocyanine Green for Detection of Endometriosis Lesions (Gre-Endo Trial): A Pilot Study.), encouraged the effort of a larger prospective trial. Based on the mini-max two-stage design by Simon [Simon R. Optimal two stage design for phase II clinical trials], the investigators tested the null hypothesis that the true rate of pathologically assessed endometriosis would improve from 87% to the clinically relevant alternative of 100.0%, as assessed by NIR-ICG laparoscopy.

DETAILED DESCRIPTION:
Patients were recruited within the clinical routine after indication for laparoscopy under consideration of the inclusion and exclusion criteria.

The sample size was calculated according to the study design by Simon (Simon R. Optimal two stage design for phase II clinical trials), using an α-error of 0.01 (two-sided) and a β-error of 0.90. Considering a patient dropout of approximately 10%, the study was planned to enrol at least 47 women.

The first abdominal and pelvi's inspection was made using direct laparoscope visualization under white light conditions. All areas suspected of peritoneal endometriosis was classified as white, black and red lesions and recorded together with their anatomic location in the surgical record for the purposes of subsequent extirpation. After the first visual inspection the patient was administered with 0.05 - 0.25 mg /(kg BW) Indocyanine Green intravenously. The Indocyanine Green imaging mode of the Olympus Indocyanine Green Imaging System was activated and suspected areas in Indocyanine Green imaging mode were recorded with them corresponding appearance in white light mode. If suspected areas were visible either in white light or Indocyanine Green imaging mode, specific sample has been taken from these areas. In addition, control biopsy specimens from inconspicuous peritoneum has been taken.

ELIGIBILITY:
Inclusion Criteria:

* Suspected endometriosis with necessity for laparoscopic confirmation and resection
* Regular menstrual cycles

Exclusion Criteria:

* Patients younger than 18 years and older than 50 years at time of operation
* Subject with previous history of adverse reaction or allergy to Indocyanine Green, iodine, shellfish or iodine dyes
* Documented allergy to sulfur containing compounds
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Indocyanine Green
* Subject has significant liver disease, cirrhosis or liver insufficiency with abnormal liver function tests (Total bilirubin increased by factor 1.5 than normal and/or serum glutamic oxaloacetic transaminase increased by factor 2 than normal)
* Subject has uremia, serum creatinine (> 2.0 mg/dl)
* Subject has severe coronary heart disease (instable angina pectoris)
* Pregnant or breast-feeding women
* Subject actively participating in another drug, biologic and/or device protocol
* The presence of medical conditions contraindicating general anesthesia or standard surgical approaches
* Subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-05-19 (Actual)

PRIMARY OUTCOMES:
Localization of occult endometriotic lesion | Intraoperative
  To detect occult endometriotic lesions, thanks to the fluorescence of the Indocyanine Green, that would remain otherwise not visible to the surgeon eye

SECONDARY OUTCOMES:
Sensibility and Specificity of Near Infrared Vision with Indocyanine green in detection of endometriotic lesions | Intraoperative
  Optical qualitative assessment through the visual evaluation of a single expert surgeon (presence / absence of fluorescence, due to the injection of the Indocyanine Green and the use of the Near Infrared vision, at the level the of suspected endometriotic lesions)
Operatory Time | Intraoperative
  To assess if the use of Indocyanine Green cause a significant increase of the operatory time
Complications | From operatory room up to 3 days
  To assess if the use of Indocyanine Green increase the percentage of intra and post-operative complications
Side effects | From operatory room up to 3 days
  Evaluation of possible side effects related to the use of Indocyanine Green as a fluorescent endometriosis' marker

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cosentino, MD, Principal Investigator — Fondazione di Ricerca e Cura Giovanni Paolo II , Campobasso , Italy
Locations (1):
- Catholic University of Sacred Heart, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cosentino F, Vizzielli G, Turco LC, Fagotti A, Cianci S, Vargiu V, Zannoni GF, Ferrandina G, Scambia G. Near-Infrared Imaging with Indocyanine Green for Detection of Endometriosis Lesions (Gre-Endo Trial): A Pilot Study. J Minim Invasive Gynecol. 2018 Nov-Dec;25(7):1249-1254. doi: 10.1016/j.jmig.2018.02.023. Epub 2018 Mar 15. PMID 29551477
- [Result] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835